CLINICAL TRIAL: NCT05726227
Title: Long-term Safety and Efficacy of Semaglutide s.c. Once-weekly on Weight Management in Children and Adolescents (Aged 6 to <18 Years) With Obesity or Overweight
Brief Title: A Research Study on How Well Semaglutide Helps Children and Teenagers With Excess Body Weight Lose Weight
Acronym: STEP Young
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4512; U1111-1266-3808 (Other: World Health Organization (WHO)); 2022-502922-41 (EudraCT Number)
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group Kids (Experimental): Participants in the age group 6 to less than (<) 12 years will receive once weekly subcutaneous (s.c.) injection of either semaglutide or placebo matched to semaglutide in dose escalation fashion for 16 weeks (0.25 mg from weeks 0-4, 0.5 mg from weeks 5-8, 1.0 mg from weeks 9-12 and 1.7 mg from weeks 13-16) followed by 2.4 mg as maintenance dose for 88 weeks as an adjunct to a reduced-calorie diet and increased physical activity.
  Interventions: Drug: Semaglutide; Drug: Placebo
- Group Teens (Experimental): Participants in the age group 12 to < 18 years will receive once weekly s.c. injection of either semaglutide or placebo matched to semaglutide in dose escalation fashion for 16 weeks (0.25 mg from weeks 0-4, 0.5 mg from weeks 5-8, 1.0 mg from weeks 9-12 and 1.7 mg from weeks 13-16) followed by 2.4 mg as maintenance dose for 88 weeks as an adjunct to a reduced-calorie diet and increased physical activity.
  Interventions: Drug: Semaglutide; Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide will be administered subcutaneously once weekly.
Drug: Placebo — Placebo will be administered subcutaneously once-weekly.

SUMMARY:
This study will look at how well semaglutide helps children and teenagers losing weight. This will be tested by comparing the effect on body weight in children and teenagers taking semaglutide in comparison to placebo, a "dummy" medicine. In addition to taking the medicine, the child's parent and the child will have talks with study staff about healthy food choices, how to be more physically active and what your child can do to try to lose weight. The child will either get semaglutide or a "dummy" medicine. Which treatment the child will get is decided by chance. Semaglutide is an approved medicine for type 2 diabetes and weight management in adults.

The child will get one injection once a week. The study medicine is injected with a thin needle in the stomach, thighs or upper arms. The study will last for about 2 ½ years (132 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of parent(s) or legally acceptable representative (LAR) of participant and child assent, as age-appropriate, obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study. a) The parents or LAR of the child must sign and date the Informed Consent Form (according to local requirements) b) The child must sign and date the Child Assent Form or provide oral assent (according to local requirements)
* Age at the time of signing informed consent. a)Group Kids: 6 to less than 12 years. b) Group Teens: 12 to less than 18 years and Tanner stage greater than 1
* Body mass index (BMI), at screening and randomisation, corresponding to a) Group Kids: greater than or equal to 95th percentile. b) Group Teens: greater than or equal to 95th percentile or greater than or equal to 85th percentile with the presence of at least 1 weight-related comorbidity (treated or untreated): hypertension, dyslipidaemia, obstructive sleep apnoea or type 2 diabetes mellitus (T2D)
* History of at least one unsuccessful effort to lose sufficient body weight after participation in a structured lifestyle modification programme (diet and exercise counselling) for at least 3 months
* Body weight of greater than 45 kilogram (kg) at screening and randomisation
* For participants with T2D at screening, the following additional criterion applies: glycated haemoglobin (HbA1c) less than or equal to 10.0 percent (86 millimoles per mole [mmol/mol]) as measured by central laboratory at screening

Exclusion Criteria:

* Treatment with any medication prescribed for the indication of obesity or weight management within 90 days before screening
* Previous or planned (during the study period) obesity treatment with surgery or a weight loss device. However, the following are allowed: a) liposuction and/or abdominoplasty, if performed greater than 1 year prior to screening. b) adjustable gastric banding, if the band has been removed greater than 1 year prior to screening. c) intragastric balloon, if the balloon has been removed greater than 1 year prior to screening. d)duodenal-jejunal bypass liner (e.g., nonbarrier), if the sleeve has been removed greater than 1 year prior to screening
* Type 1 diabetes mellitus or monogenic diabetes
* Participants with endocrine, hypothalamic, or syndromic obesity
* For participants with T2D at screening, the following additional key criterion applies: Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
Group Kids: Change in body mass index (BMI) | From baseline (week 0) to week 68
  Measured in percentage (%)

SECONDARY OUTCOMES:
Group Kids: Improvement in weight category | From baseline (week 0) to week 68
  Measured as count of participants. Weight categories based on growth charts from Center for Disease Control (CDC).gov: Normal weight= BMI less than (<) 85th percentile, Overweight= BMI greater than or equal to (>=) 85th - <95th percentile, Obesity class I= BMI >=95th - <120% of the 95th percentile, Obesity class II= BMI >=120% - <140% of the 95th percentile, Obesity class III= BMI >=140% of the 95th percentile.
Group Teens: Change in BMI | From week 0 to week 68
  Measured in %
Group Kids and Group Teens: Change in BMI | From week 0 to week 104
  Measured in %
Group Teens: Improvement in weight category | From week 0 to week 68
  Measured as count of participants. Weight categories based on growth charts from CDC.gov: Normal weight= BMI less than (<) 85th percentile, Overweight= BMI greater than or equal to (>=) 85th - <95th percentile, Obesity class I= BMI >=95th - <120% of the 95th percentile, Obesity class II= BMI >=120% - <140% of the 95th percentile, Obesity class III= BMI >=140% of the 95th percentile.
Group Kids and Group Teens: Improvement in weight category | From week 0 to week 104
  Measured as count of participants. Weight categories based on growth charts from CDC.gov: Normal weight= BMI less than (<) 85th percentile, Overweight= BMI greater than or equal to (>=) 85th - <95th percentile, Obesity class I= BMI >=95th - <120% of the 95th percentile, Obesity class II= BMI >=120% - <140% of the 95th percentile, Obesity class III= BMI >=140% of the 95th percentile.
Group Kids and Group Teens: Change in body weight | From week 0 to week 68
  Measured in percentage
Group Kids and Group Teens: Change in body weight | From week 0 to week 104
  Measured in percentage
Group Kids and Group Teens: Change in body weight | From week 0 to week 68
  Measured in kilograms (kg)
Group Kids and Group Teens: Change in body weight | From week 0 to week 104
  Measured in kilograms (kg)
Group Kids and Group Teens: Change in BMI percentage of the 95th percentile | From week 0 to week 68
  Measured in percentage points
Group Kids and Group Teens: Change in BMI percentage of the 95th percentile | From week 0 to week 104
  Measured in percentage points
Group Kids and Group Teens: Change in BMI Standard deviation score (SDS) | From week 0 to week 68
  Measured as score on a scale. BMI SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' BMI provided for each sex and age. For each subject, a Z (SDS) score was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction.
Group Kids and Group Teens: Change in BMI SDS | From week 0 to week 104
  Measured as score in a scale. BMI SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' BMI provided for each sex and age. For each subject, a Z (SDS) score was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction.
Group Kids and Group Teens: Change in waist circumference | From week 0 to week 68
  Measured in centimeters (cm)
Group Kids and Group Teens: Change in waist circumference | From week 0 to week 104
  Measured in centimeters (cm)
Group Kids and Group Teens: Change in systolic blood pressure | From week 0 to week 68
  Measured in millimeters of mercury (mmHg)
Group Kids and Group Teens: Change in systolic blood pressure | From week 0 to week 104
  Measured in millimeters of mercury (mmHg)
Group Kids and Group Teens: Change in diastolic blood pressure | From week 0 to week 68
  Measured in mmHg
Group Kids and Group Teens: Change in diastolic blood pressure | From week 0 to week 104
  Measured in mmHg
Group Kids and Group Teens: Change in total cholesterol | From week 0 to week 68
  Measured in %
Group Kids and Group Teens: Change in total cholesterol | From week 0 to week 104
  Measured in %
Group Kids and Group Teens: Change in high density lipoprotein (HDL) | From week 0 to week 68
  Measured in %
Group Kids and Group Teens: Change in high density lipoprotein (HDL) | From week 0 to week 104
  Measured in %
Group Kids and Group Teens: Change in low density lipoprotein (LDL) | From week 0 to week 68
  Measured in %
Group Kids and Group Teens: Change in low density lipoprotein (LDL) | From week 0 to week 104
  Measured in %
Group Kids and Group Teens: Change in very low density lipoprotein (VLDL) | From week 0 to week 68
  Measured in %
Group Kids and Group Teens: Change in very low density lipoprotein (VLDL) | From week 0 to week 104
  Measured in %
Group Kids and Group Teens: Change in triglycerides | From week 0 to week 68
  Measured in %
Group Kids and Group Teens: Change in triglycerides | From week 0 to week 104
  Measured in %
Group Kids and Group Teens: Change in high sensitivity C-reactive protein (hs-CRP) | From week 0 to week 68
  Measured in %
Group Kids and Group Teens: Change in high sensitivity C-reactive protein (hs-CRP) | From week 0 to week 104
  Measured in %
Group Kids and Group Teens: Change in glycated haemoglobin (HbA1c) | From week 0 to week 68
  Measured in % point
Group Kids and Group Teens: Change in glycated haemoglobin (HbA1c) | From week 0 to week 104
  Measured in % point
Group Kids and Group Teens: Change in fasting plasma glucose | From week 0 to week 68
  Measured in millimoles per liter (mmol/L)
Group Kids and Group Teens: Change in fasting plasma glucose | From week 0 to week 104
  Measured in millimoles per liter (mmol/L)
Group Kids and Group Teens: Change in fasting plasma glucose | From week 0 to week 68
  Measured in milligrams per deciliter (mg/dL)
Group Kids and Group Teens: Change in fasting plasma glucose | From week 0 to week 104
  Measured in milligrams per deciliter (mg/dL)
Group Kids and Group Teens: Change in fasting insulin | From week 0 to week 68
  Measured in %
Group Kids and Group Teens: Change in fasting insulin | From week 0 to week 104
  Measured in %
Group Kids and Group Teens: Change in alanine transaminase (ALT) | From week 0 to week 68
  Measured in milliunits per liter (mU/L)
Group Kids and Group Teens: Change in alanine transaminase (ALT) | From week 0 to week 104
  Measured in milliunits per liter (mU/L)
Group Kids and Group Teens: Change in total fat mass, by Dual energy X-ray absorptiometry (DXA) relative to total body mass | From week 0 to week 68
  Measured in % points
Group Kids and Group Teens: Change in total fat mass, by Dual energy X-ray absorptiometry (DXA) relative to total body mass | From week 0 to week 104
  Measured in % points
Group Kids and Group Teens: Change in lean body mass, by DXA relative to total body mass | From week 0 to week 68
  Measured in % points
Group Kids and Group Teens: Change in lean body mass, by DXA relative to total body mass | From week 0 to week 104
  Measured in % points
Group Kids and Group Teens: Relative change in visceral fat mass by DXA | From week 0 to week 68
  Measured in %
Group Kids and Group Teens: Relative change in visceral fat mass by DXA | From week 0 to week 104
  Measured in %
Group Kids and Group Teens: Number of participants achieving greater than or equal to (>=) 5% reduction of BMI (yes/no) | From week 0 to week 68
  Measured in count of participants
Group Kids and Group Teens: Number of participants achieving greater than or equal to (>=) 5% reduction of BMI (yes/no) | From week 0 to week 104
  Measured in count of participants
Group Kids and Group Teens: Number of participants achieving greater than or equal to (>=) 10% reduction of BMI (yes/no) | From week 0 to week 68
  Measured in count of participants
Group Kids and Group Teens: Number of participants achieving greater than or equal to (>=) 10% reduction of BMI (yes/no) | From week 0 to week 104
  Measured in count of participants
Group Kids and Group Teens: Number of participants achieving greater than or equal to (>=) 15% reduction of BMI (yes/no) | From week 0 to week 68
  Measured in count of participants
Group Kids and Group Teens: Number of participants achieving greater than or equal to (>=) 15% reduction of BMI (yes/no) | From week 0 to week 104
  Measured in count of participants
Group Kids and Group Teens: Number of treatment emergent adverse events (AEs) | From week 0 to week 68
  Measured as count of events
Group Kids and Group Teens: Number of treatment emergent adverse events (AEs) | From week 0 to week 111
  Measured as count of events
Group Kids and Group Teens: Number of treatment emergent serious adverse events (SAEs) | From week 0 to week 68
  Measured as count of events
Group Kids and Group Teens: Number of treatment emergent serious adverse events (SAEs) | From week 0 to week 111
  Measured as count of events
Group Kids and Group Teens: Change in pulse | From week 0 to week 68
  Measured as beats per minute
Group Kids and Group Teens: Change in pulse | From week 0 to week 104
  Measured as beats per minute
Group Kids and Group Teens: Change in amylase | From week 0 to week 68
  Measured as units per liter (U/L)
Group Kids and Group Teens: Change in amylase | From week 0 to week 104
  Measured as units per liter (U/L)
Group Kids and Group Teens: Change in lipase | From week 0 to week 68
  Measured as U/L
Group Kids and Group Teens: Change in lipase | From week 0 to week 104
  Measured as U/L
Group Kids and Group Teens: Change in calcitonin | From week 0 to week 68
  Measured as nanograms per liter (ng/L)
Group Kids and Group Teens: Change in calcitonin | From week 0 to week 104
  Measured as nanograms per liter (ng/L)
Group Kids and Group Teens: Change in bone mineral density, by DXA | From week 0 to week 68
  Measured as grams per square centimeter (g/cm^2)
Group Kids and Group Teens: Change in bone mineral density, by DXA | From week 0 to week 104
  Measured as grams per square centimeter (g/cm^2)
Group Kids and Group Teens: Number of treatment emergent hypoglycaemic episodes (for T2D only) | From week 0 to week 68
  Measured as count of episodes
Group Kids and Group Teens: Number of treatment emergent hypoglycaemic episodes (for T2D only) | From week 0 to week 111
  Measured as count of episodes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (56):
- United States (24):
  - Neighborhood Healthcare, Escondido, California
  - Yale School of Medicine, New Haven, Connecticut
  - Columbus Research Foundation, Columbus, Georgia
  - Eastside Bariatric and Gen Surg, Snellville, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Pennington Biom Res Ctr, Baton Rouge, Louisiana
  - Clinical Trials of America LLC, Monroe, Louisiana
  - IMA Clinical Research, Monroe, Louisiana
  - Barry J. Reiner, MD LLC, Baltimore, Maryland
  - Massachusetts General Hospital_Cary, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Mississippi CTR for ADV MED, Madison, Mississippi
  - UBMD Peds-Div of Endo/Diabetes, Buffalo, New York
  - WakeMed Childn Endo-Dbt_Raleig, Raleigh, North Carolina
  - Valley Weight Loss Clinic, Fargo, North Dakota
  - Centricity Research - Ohio, Columbus, Ohio
  - UPMC Child Hosp-Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Tullahoma Pediatrics PLLC, Tullahoma, Tennessee
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Univ Of Texas Hlth Science Cntr, San Antonio, Texas
  - Health Res of Hampton Roads, Newport News, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Austria (2):
  - Universitätsklinik Kinder-Jugendheilkunde Innsbruck, Innsbruck
  - Universitätsklinik für Kinder und Jugendheilkunde Haus E, Salzburg
- Belgium (4):
  - UZ Brussel, Brussels
  - UZ Antwerpen - UZA - Kinderziekenhuis, Edegem
  - UZA - UZ Antwerpen - Kinderziekenhuis, Edegem
  - UZ Leuven - Kindergeneeskunde, Leuven
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Steno Diabetes Center Aarhus, Aarhus
  - Holbæk Sygehus - Børne- og Ungeafdelingen, Holbæk
- Germany (7):
  - Universitätsklinikum Halle - Innere Medizin II, Halle
  - Hannoversche Kinderheilanstalt "Auf der Bult" - Diabeto-, Endokrino-, Gastroenterologie und Klinische Forschung, Hanover
  - Kinder- und Jugendkrankenhaus, Hanover
  - Uniklinik Leipzig - Klinik und Poliklinik für Kinder- und Jugendmedizin, Leipzig
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Kinder- und Jugendmedizin, Leipzig
  - Uniklinik Ulm - Dt. Zentrum für Kinder- und Jugendgesundheit (DZKJ), Ulm
  - Universitätsklinikum Ulm für Kinder- und Jugendmedizin, Ulm
- Israel (3):
  - Rambam MC - Department of Pediatrics A, Haifa
  - Schneider MC - Endrocrinology and Diabetes, Petah Tikva
  - Shamir MC - Pediatric and Adolescents Endocrinology unit, Ẕerifin
- Consultorio de Endocrinología y Pediatría, Puebla City, Mexico
- Portugal (3):
  - Hospital Da Luz S.A., Lisbon
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
  - Hospital CUF Porto S.A., Porto
- Sweden (4):
  - Drottning Silvias barnsjukhus, Gothenburg
  - Hallands sjukhus Halmstad, Halmstad
  - Akademiska sjukhuset Uppsala, Uppsala
  - Uppsala universitetssjukhus, Uppsala
- United Kingdom (5):
  - Birmingham Children's Hospital, Birmingham
  - University Hospitals Bristol & Weston NHS Foundation Trust, Bristol
  - Leeds Children's Hospital, Leeds
  - Alder Hey Children's Hospital, Liverpool
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com